CLINICAL TRIAL: NCT06110962
Title: Detecting Heart Rate, Respiration, and Sleep With the Sleeptracker-AI Under-mattress Monitor
Status: Recruiting | Type: Observational
Sponsor: Woolcock Institute of Medical Research (Other)
Collaborators: Fullpower Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: X23-0255
Record Dates: First submitted 2023-10-24; First posted 2023-11-01 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: OSA
Keywords: validation study; Sleeptracker-AI; polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients: Sleep clinic patients undergoing polysomnography sleep studies for diagnosis of sleep apnea
  Interventions: Device: Sleeptracker-AI

INTERVENTIONS:
Device: Sleeptracker-AI — The Sleeptracker-AI Monitor (Fullpower Technologies, California, USA) is a commercially available, unobtrusive, and non-wearable home sleep monitoring device. It is either pre-installed in a mattress or can be purchased separately by consumers where it is placed under the mattress. The device uses piezo-electric sensors that register the forces exerted through the mattress by features such as the subject's motion, respiration, heartbeats, and snoring vibrations.

SUMMARY:
The objective of this study is to simultaneously acquire sleep and breathing data using the under-mattress Sleeptracker (The Sleeptracker-AI Monitor (Fullpower Technologies, California, USA) during routine PSGs in patients who attend the Woolcock Institute for undergoing investigation for possible obstructive sleep apnoea (OSA).

DETAILED DESCRIPTION:
The objective of this study is to simultaneously acquire sleep and breathing data using the under-mattress Sleeptracker (The Sleeptracker-AI Monitor (Fullpower Technologies, California, USA) during routine PSGs in patients who attend the Woolcock Institute for undergoing investigation for possible obstructive sleep apnoea (OSA). The de-identified Sleeptracker and PSG data will then be used by Fullpower Technologies to improve the accuracy of their current algorithm for detecting sleep and breathing disorders using the Sleeptracker device.

De-identified data recorded from the Sleeptracker device and PSG data from the Compumedics Grael system will be manually uploaded to a secure commercial server maintained by Fullpower Technologies.

Fullpower Technologies will use the de-identified data to refine their algorithms for detecting sleep and breathing disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-90 years old at time of assessment.
* Attending the Woolcock Institute for an overnight sleep study for investigation of sleep apnoea.
* Able to give informed consent.
* Fluent in English.

Exclusion Criteria:

* Unable to understand study procedure.
* Unable to sign informed consent form.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Woolcock Institute for a diagnostic sleep study for possible sleep apnea.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2028-10-10 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | One night
  AHI (events per hour of sleep)

SECONDARY OUTCOMES:
Total Sleep Time | One night
  Total Sleep Time (minutes)
NREM Sleep Time | One night
  Non-REM sleep time (minutes)
REM Sleep Time | One night
  REM sleep time (minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Phillips, PhD, Principal Investigator — Woolcock Institute of Medical Research
Locations (1):
- Woolcock Institute of Medical Research, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Data collected during the study are completed de-identifiable and will be sent to FullPower for algorithm training purposes. No identifiable data will be shared.